CLINICAL TRIAL: NCT01630785
Title: Retrospective Data Analysis of Neurophysiological Data for Intraoperative or Epilepsy Monitoring
Brief Title: Neurophysiological Intraoperative or Epilepsy Monitoring
Acronym: nphysdocu
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: nphysdocu
Record Dates: First submitted 2012-06-21; First posted 2012-06-28 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Patients Operated on at the Neurosurgery Department
MeSH Terms: interventions — Intraoperative Neurophysiological Monitoring

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years

GROUPS / COHORTS (1):
- IONM patients: all patients where surgery requires IONM
  Interventions: Device: Intraoperative Neurophysiological Monitoring IONM

INTERVENTIONS:
Device: Intraoperative Neurophysiological Monitoring IONM — Intraoperative Neurophysiological Monitoring IONM device. Manufacturer: Inomed, Emmendingen, Germany

SUMMARY:
The investigators record the outcome of patients whose surgery involved intraoperative neurophysiological monitoring

* Trial with surgical intervention

ELIGIBILITY:
Inclusion criteria: Patients whose surgery involved intraoperative neurophysiological monitoring

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients whose surgery involved intraoperative neurophysiological monitoring
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2012-01; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
oncological outcome | 5 years
  overall survival, progression free survival
neurological outcome | 1 year
  validated scales like Karnofsky or NIHSS
seizure outcome | 1 year
  ILAE classification of epilepsy surgery outcome

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Sarnthein, Prof Dr, Principal Investigator — University Hospital Zurich, Division of Neurosurgery; Oliver Bozinov, PD Dr, Principal Investigator — University Hospital Zurich, Division of Neurosurgery; Niklaus Krayenbühl, Prof Dr, Principal Investigator — University Hospital Zurich, Division of Neurosurgery; Luca Regli, Prof Dr, Principal Investigator — University Hospital Zurich, Division of Neurosurgery
Locations (1):
- University Hospital Zurich, Neurosurgery, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Yang Y, Neidert MC, Velz J, Kalin V, Sarnthein J, Regli L, Bozinov O. Mapping and Monitoring of the Corticospinal Tract by Direct Brainstem Stimulation. Neurosurgery. 2022 Sep 1;91(3):496-504. doi: 10.1227/neu.0000000000002065. Epub 2022 Jul 14. PMID 35876678